CLINICAL TRIAL: NCT06535802
Title: iCCaRE Consortium Pilot Project 1: Feasibility of a Point of Prostate Cancer Diagnosis Intervention for Newly Diagnosed Black Men
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MC220501; W81XWH2210968 (Other Grant/Funding Number: Department of Defense); NCI-2024-05156 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC220501 (Other: Mayo Clinic in Florida); 22-001412 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Observational cohort I: Consumer advocates attend a focus group on study.
  Interventions: Other: Focus group
- Observational cohort II: Clinicians complete interviews on study.
  Interventions: Other: Clinician Interviews
- Observational cohort III: CaP survivors test the virtual health intervention, complete a survey, and attend a focus group on study.
  Interventions: Other: Focus group; Other: Intervention testing; Other: Survey
- Observational cohort V: Patients complete surveys and participate in the virtual health intervention on study. Patients complete survey and an interview during follow up.
  Interventions: Other: Survey; Other: Follow-up Interview; Other: Virtual Health Intervention

INTERVENTIONS:
Other: Focus group — Attend a focus group session
  Groups: Observational cohort I; Observational cohort III
Other: Clinician Interviews — Participate in clinician interviews
  Groups: Observational cohort II
Other: Intervention testing — Test the virtual health intervention
  Groups: Observational cohort III
Other: Survey — Complete a follow-up survey
  Groups: Observational cohort III; Observational cohort V
Other: Follow-up Interview — Participate in a follow-up interview
  Groups: Observational cohort V
Other: Virtual Health Intervention — Participate in the virtual health intervention
  Groups: Observational cohort V

SUMMARY:
This study is being done to determine the acceptance and effectiveness of a virtual robot assistant model at a urology clinic.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Plan and develop a PPCD iCCaRE ViRA model that will provide social determinants of health (SDOH) navigation services, psycho-oncology support and emotional support using qualitative formative research.

II: Establish the acceptance and usability of the iCCaRE ViRA among 50 African American/Black men (AA/BM) at local Jacksonville sites.

OUTLINE: This is an observational study. Participants are assigned to 1 of 4 cohorts.

COHORT I: Consumer advocates attend a focus group on study.

COHORT II: Clinicians complete interviews on study.

COHORT III: CaP survivors test the virtual health intervention, complete a survey, and attend a focus group on study.

COHORT IV: Patients complete surveys and participate in the virtual health intervention on study. Patients complete survey and an interview during follow up.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: iCCaRE Consortium consumer advocates
* Clinicians who are part of the Translational Research & Clinical Intervention Services (TRaCIS)
* AIM 2 ALPHA TESTING: iCCaRE consumer advocates [2 Community Advisory Board (CAB) and 1 non-CAB]
* AIM 2 BETA TESTING-PATIENTS:

  * An African American/Black male
  * A patient who has been diagnosed with prostate cancer in Florida at any time in their life, and/or within the previous 6 months has had an abnormal Prostate-Specific Antigen (PSA) lab value and/or Digital Rectal Examination (DRE)
  * Minimum age of 30 years old
  * Consent to participating in the intervention

Exclusion Criteria:

* AIM 2 BETA TESTING-PATIENTS:

  * Patients who are not African American/Black males
  * Patients not diagnosed with prostate cancer in Florida at any time in their life, or within the previous 6 months has not had a normal PSA lab value and/or DRE
  * Older than 80 years old
  * Are not willing to consent

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: iCCaRE Consortium consumer advocates, clinicians as part of the iCCaRE Consortium Translational Research & Clinical Intervention Services. Community Advisory Board (CAB) and non-CAB iCCaRE consumer advocates. Patients with an abnormal PSA and/or DRE diagnosed with prostate cancer in the state of Florida.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Point of Prostate Cancer Diagnosis (PPCD) iCCaRE Virtual Reality Assistant (ViRA) model | Up to 4 months
  Will be assessed by the length of time needed to create the model. PPCD iCCaRE ViRA model development will be guided by the Translational Research & Clinical Intervention Services (TRaCIS) and Digital Health & Human Services (DHHS) core sections of the Inclusive Cancer Care Research Equity (iCCaRE) Consortium. The consortium's scientific team and Community Advisory Board (CAB) will participate in making decisions about how to proceed with the development of the ViRA Intervention and Communication Strategy Plan (ICoSP). This application (app) will be evaluated in Outcomes 2 and 3. The PPCD iCCaRE ViRA app will provide social determinants of health (SDOH) navigation services, psycho-oncology support and emotional support using qualitative formative research.
Acceptance of the iCCaRE ViRA | Baseline; follow-up interview 3-4 months post visit
  Will be assessed by patient immediate reaction and patient delayed feedback.
Usability of the iCCaRE ViRA | Baseline; follow-up interview 3-4 months post visit
  Will be assessed by patient immediate reaction and patient delayed feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Folakemi T. Odedina, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials